CLINICAL TRIAL: NCT02468297
Title: Efficacy of the Electronic Acupuncture Shoes: A Clinical Trial for Chronic Low Back Pain
Acronym: EAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Yu Sheng (Other)
Responsible Party: Sponsor-Investigator, Chen Yu Sheng, Medical Doctor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 92-0530A
Record Dates: First submitted 2015-06-06; First posted 2015-06-10 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Electronic Acupuncture Shoe (Experimental): Experiment group receives a one-hour treatment given by "Electronic Acupuncture Shoe" three times a week. 6 weeks of treatment was given. Subjects took placebo only in the first week. No placebo or medicine was prescribed to the subjects since the second week.
  Interventions: Device: Electronic Acupunture Shoes
- Control group (Placebo Comparator): Control group received the six-week treatment as well, yet the subjects received pseudo electrotherapy. Subjects took ibuprofen(400mg, TID) only in the first week. No placebo or medicine was prescribed to the subjects since the second week.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Device: Electronic Acupunture Shoes — Experiment group receives a one-hour treatment given by "Electronic Acupuncture Shoes" three times a week. 6 weeks of treatment was given.
  Control group received the six-week treatment as well, yet the subjects received pseudo electrotherapy.
  Arms: Electronic Acupuncture Shoe
Drug: Ibuprofen — Experiment group took placebo only in the first week. Control group took ibuprofen(400mg, TID) only in the first week. No more placebo or medicine was prescribed to either two groups since the second week.
  Arms: Control group

SUMMARY:
This randomized , double-blind, parallel-arm clinical trial was designed to study the efficacy and safety of the "Electronic Acupuncture Shoes" treatment on chronic low back pain patients.

Chronic low back pain patients, aged 20-60, of both gender were recruited. As the primary outcome measure to assess the efficacy, "0-10 numerical rating scale" was used. Secondary outcome measure included the speed of pain-relief.

The number of samples in the experimental group and the control group ratio of 1 : 1 , is expected to total effective sample number is 60 . Experimental group will receive a six-week "Electronic Acupuncture Shoes" treatment and a week back to the clinic three times , subject to a total of 18 treatments , each course of about one hour . Subjects will take NSAID placebo in the first week of the course of treatment . After the second week of NSAID placebo on disabled.

Control subjects will also accept the six- week treatment , control subjects will be equally back to the clinic three times a week , each group will be given to the subject of one hour each shoe pseudo electrotherapy treatment group and control group run by entering from the test day in the first week of the course , each taking ibuprofen 400mg, taken three times a day , the second week after the NSAID drugs on disabled.

ELIGIBILITY:
Inclusion Criteria:

A. Diagnosed with chronic low back pain (pain that persists for more than 12 weeks ).

B. Subjects who agreed to be involved and signed the agreement, after being explained to by the investigators.

Exclusion Criteria:

A. Diagnosed with cancer . B. Early menopause ( before age 50 ) . C. Ovariectomized D. Under steroid therapy E. Rheumatoid arthritis F. With fractures or have undergone back surgery. G. Compression syndrome: e.g. HIVD ( Herniated Intervertebral Disc) , spinal disorder .

H. Renal calculus. I. Pacemaker users . J. Pregnant women or women who expect to be pregnant. K. Visual impairment . L. Diabetes. M. Visceral infections, e.g. pancreatitis, nephritis . N. Under other clinical trials (under medication or given other treatment) within 30 days before . O. Contraindications of ibuprofen. P. Poor function of heart, liver, GI tract or kidney. Q. Be suspected by the doctors of potential illness, disease or any other reason, which may endanger the subjects .

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-04-15 (Actual); Primary Completion 2012-01-30 (Actual); Study Completion 2012-01-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 6 weeks

SECONDARY OUTCOMES:
The speed of pain-relief | 6 weeks

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeh BY, Liu GH, Lee TY, Wong AM, Chang HH, Chen YS. Efficacy of Electronic Acupuncture Shoes for Chronic Low Back Pain: Double-Blinded Randomized Controlled Trial. J Med Internet Res. 2020 Oct 26;22(10):e22324. doi: 10.2196/22324. PMID 33104004